CLINICAL TRIAL: NCT03331016
Title: Evaluating the Effectiveness of a Sexual Health Curriculum for Foster and Kinship Caregivers
Brief Title: Heart to Heart: Testing a Sexual Health Training for Foster and Kinship Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Kym Ahrens, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-022514-S
Record Dates: First submitted 2017-10-06; First posted 2017-11-06 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Sexual Behavior; Conflict, Family; Pregnancy Related; Sexually Transmitted Diseases; Family and Household
Keywords: Foster caregiver; Kinship caregiver; Foster youth; Unintended pregnancy; Curriculum; Intervention; sexually transmitted infections; Behaviorism; Monitoring; Communication; Adolescent development; sexually transmitted diseases
MeSH Terms: conditions — Sexual Behavior; Sexually Transmitted Diseases; Communication

STUDY DESIGN:
Intervention Model Description: Randomized stepped wedge design with waitlist controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control Group (Other): Waitlist Control Group will serve as control group for 6 months, receiving no intervention during that time but completing periodic surveys to assess outcomes among controls (knowledge, attitudes, behaviors). They will also later receive the intervention (training program) and be followed for 6 more months.
  Interventions: Behavioral: Heart to Heart Training
- Intervention Group (Experimental): Intervention Group will receive the intervention (training program) right away, then will be followed for 6 months.
  Interventions: Behavioral: Heart to Heart Training

INTERVENTIONS:
Behavioral: Heart to Heart Training — Training for foster and kinship caregivers on sexual health and how to effectively communicate with and monitor youth in their care, with the aim of reducing unintended pregnancies and sexually transmitted infections in this youth population.

SUMMARY:
Heart to Heart is a brief pregnancy prevention training program delivered to foster and kinship caregivers to prevent unintended pregnancy in foster youth. The training delivers easy to understand information on sexual health, contraception, and adolescent development. It also includes a brief behavioral training, and information on effective communication, monitoring strategies, and social support. The curriculum was piloted in Los Angeles. Investigators will test the intervention in a randomized control trial.

DETAILED DESCRIPTION:
Dr. Ahrens and her team will evaluate the effectiveness of this training using a randomized stepped wedge study design with a target enrollment of 100 foster and kinship caregivers. Recruitment will be carried out in collaboration with the Los Angeles Department of Child and Family Services, foster family agencies and support groups. After completing a baseline survey, participants will be randomly assigned to either the intervention group or the waitlist control group. (With a target 1:1 ratio of controls to intervention subjects, but in consideration of greater levels of attrition in the waitlist control group due to the 6-month wait before being offered the training, participants will be randomized in a ratio of 4:3 to control vs intervention group). The intervention group will receive the training soon after enrollment, and will then complete 3 follow-up surveys over the following 6 months. Participants assigned to the waitlist control group will first complete 3 surveys over 6 months, receive the intervention at the 6 month mark, then take 3 follow-up surveys over the following 6-month period. Dr. Ahrens and team will use these survey data to measure the effectiveness of the training based on the outcome measures. Participants will be surveyed at multiple timepoints both because the different outcomes are expected to occur within different time intervals (e.g. knowledge may change right away, while behaviors will take longer), and to assess whether these outcomes change over time (e.g. whether knowledge gained in the training is lasting).

ELIGIBILITY:
Inclusion Criteria:

* Is a foster or kinship caregiver in Los Angeles County.
* Has a youth age 11-21 who has lived with them for at least 3 months in the past year.
* Anticipates that at least one youth age 11-21 will continue to live with them for the next 12 months.
* Is available for either training group (immediate or in 6 months).

Exclusion Criteria:

* Does not anticipate youth will stay in their home for 12 months
* Does not have a youth age 11-21 in their home
* Cannot commit to being randomized to either training group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Sexual Health Knowledge Scale (adapted from Sexual Knowledge and Attitude Test for Adolescents by Fullard, Scheier, & Lief, 2005) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Assessing caregivers' basic knowledge about sexual health via Sexual Knowledge and Attitude Test for Adolescents measure. Total score range = 0-8, higher = better.
Parental Monitoring Scale (Stattin & Kerr, 2000) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Assessing the degree to which caregivers are aware of youth's whereabouts and activities. Total score range = 5-25, higher = better.
Parenting Outcome Expectancy Scale | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Change in parent expectations about discussing sexual health topics over time. Total score range = 6-30, higher = better.
Conflict Behavior Questionnaire (Robin & Foster, 1989) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Assessing amount of conflict between caregiver and foster youth. Total score range = 20-80, higher = better.
Media Communication and Monitoring (non-validated scale) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Change in media discussions and monitoring behaviors - 2 question questionnaire developed by Megan Moreno questions available upon request. Total score range = 5-10, higher = better)
Barriers to Talking about Sex (non-validated scale) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Change in number of barriers to caregivers talking about sex with teens in their home. Questionnaire developed by research team based on focus group data.
Sexual Communication Behaviors Scale (adapted from Dutra, Miller, Forehand, 1999) | We will assess change from baseline over 6 months in each arm (outcomes will be measured at baseline, 1 month, 3 months, and 6 months).
  Change in number of sexual health topics discussed with youth and how helpful caregivers perceive conversations to be. Total score range = 0-11, lower = better); 3 subscales: 1) Number of topics = 0-6, higher = better; 2) Frequency of communication = 0-4, higher = better; 3) Helpfulness of conversations = 1-3, higher = better.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pasadena City College, Pasadena, California
  - Los Angeles Mission College, Sylmar, California

IPD SHARING:
Plan to Share IPD: No
The investigators do not have specific plans to make IPD available to other researchers, but they are open to it if there is interest from other investigators.

REFERENCES:
- [Derived] Ahrens KR, Udell W, Albertson K, Lowry S, Hoopes T, Coatney A. Development and two-phased pilot RCT of a foster/kinship caregiver intervention to improve sexual health communication with youth. Child Youth Serv Rev. 2021 Mar;122:105877. doi: 10.1016/j.childyouth.2020.105877. Epub 2020 Dec 25. PMID 34992327